CLINICAL TRIAL: NCT03049280
Title: A Prospective, Multicenter Investigation of the da Vinci® SP™ Surgical System in TORS Procedures for Resection of Malignant Tumors
Brief Title: Prospective, Multicenter da Vinci® SP™ Surgical System TORS Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISI dV SP-TORS - 01
Record Dates: First submitted 2017-01-30; First posted 2017-02-10 (Actual); Results first posted 2020-08-18 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Oropharyngeal Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Transoral robotic surgery (Experimental)
  Interventions: Device: Transoral robotic surgery

INTERVENTIONS:
Device: Transoral robotic surgery — Transoral robotic surgery for T1 & T2 oropharyngeal cancers

SUMMARY:
A prospective, multicenter investigation of the da Vinci® SP™ Surgical System in Transoral Robotic Surgery (TORS) procedures for malignant oropharyngeal tumors.

DETAILED DESCRIPTION:
A prospective, multicenter investigation to evaluate the safety and clinical performance of the da Vinci SP Surgical System, instruments, and accessories in TORS procedures for malignant oropharyngeal tumors classified as T1 and T2.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* T1 or T2 malignant oropharyngeal tumor
* Tumor amenable to transoral resection
* No previous treatment for the index tumor
* Willing and able to provide written informed consent
* Willing and able to comply with the study protocol requirements

Exclusion Criteria:

* T3 or T4 stage tumor
* Previous radiation treatment to the head and neck, with or without chemotherapy
* Evidence of other primary cancers or distant metastasis or subject with synchronous primary tumor excluding skin cancers
* Pre-operative expectation of needing microvascular soft-tissue reconstruction
* Tumor that invades and/or abuts the internal and/or external carotid artery
* Retropharyngeal carotid artery coincident with a tonsillar cancer or posterior pharyngeal wall cancer
* Evidence of mandibular invasion of tumor
* Eastern Cooperative Oncology Group Performance Status score greater than or equal to 2
* On a medication that interferes with clotting that cannot be stopped prior to surgery
* Contraindication for general anesthesia or surgery
* Mentally handicapped or has psychological disorder or severe systemic illness that would preclude compliance with study requirements or ability to provide informed consent
* Pregnant or suspected to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Holsinger, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Board of Trustees of the Leland Stanford Junior University, Palo Alto, California
  - Florida Hospital, Celebration, Florida
  - Trustees of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holsinger FC, Magnuson JS, Weinstein GS, Chan JYK, Starmer HM, Tsang RKY, Wong EWY, Rassekh CH, Bedi N, Hong SSY, Orosco R, O'Malley BW Jr, Moore EJ. A Next-Generation Single-Port Robotic Surgical System for Transoral Robotic Surgery: Results From Prospective Nonrandomized Clinical Trials. JAMA Otolaryngol Head Neck Surg. 2019 Nov 1;145(11):1027-1034. doi: 10.1001/jamaoto.2019.2654. PMID 31536129

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of study subjects occurred between April 2017 and October 2017 at 3 participating sites
Groups:
- TORS: Subjects that underwent transoral otolaryngology robotic surgery
Period: Overall Study
Arm/Group | TORS
Started | 33
Completed | 32
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Subjects were evaluated for eligibility into the study using medical history, medical exam and imaging
Arm/Group | TORS
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 30
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Performance
Description: Performance defined as the conversion to an open approach required to complete the procedure
Time Frame: Intraoperative
Population: all subjects that were eligible to participate and underwent TORS
Measure: Count of Participants; unit: Participants
Groups:
- TORS: subjects undergoing transoral otolaryngology robotic surgery
Arm/Group | TORS
Number analyzed (Participants) | 33
Participants | 0

2. Primary Outcome: Number of Subjects With Device-related Serious Adverse Events
Description: Safety is determined by measuring the number of subjects that experience device-related serious adverse events
Time Frame: Intraoperative period
Population: Subject that were eligible to participate and underwent TORS
Measure: Count of Participants; unit: Participants
Arm/Group | TORS
Number analyzed (Participants) | 33
Participants | 0

3. Secondary Outcome: Positive Surgical Margin
Description: Rate of final positive surgical margins confirmed by pathology
Time Frame: Through14-days postoperatively
Measure: Count of Participants; unit: Participants
Groups:
- TORS: Subject undergoing transoral otolaryngology robotic surgery
Arm/Group | TORS
Number analyzed (Participants) | 33
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the conduct of the study and through 7 weeks follow-up
Arm/Group | TORS
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 4/33
Other Adverse Events (participants affected / at risk) | 4/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TORS (N=33)
Hypoxemia (General disorders) | 1 (1)
Left middle cerebral artery (MCA) stroke (Vascular disorders) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hospital-acquired
clostridium difficile enterocolitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TORS (N=33)
Neck seroma (Skin and subcutaneous tissue disorders) | 1 (1)
Nasal regurgitation (General disorders) | 1 (1)
Fall (Social circumstances) | 1 (1)
Trismus (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT03049280/Prot_SAP_000.pdf